CLINICAL TRIAL: NCT05696132
Title: Evaluation of the Decolonization Rate and Acceptance of a Complete Nasal Decolonization Kit With Povidone Iodine for MRSA Patients
Acronym: MRSAD-PVP-I
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC21_0556
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: MRSA
MeSH Terms: interventions — Povidone-Iodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decolonization (Experimental): Nasal decolonization with betadin gel
  Interventions: Drug: Betadine

INTERVENTIONS:
Drug: Betadine — Nasal decolonization with betadine gel

SUMMARY:
Staphylococcus aureus (S. aureus) is a leading cause of healthcare-associated infections worldwide. S. aureus colonizes several body sites, including the nose, throat, and perineum. Colonization by methicillin-resistant S. aureus (MRSA) increases the risk of infection by up to 27%, with infecting strains matching colonizing strains in up to 86% of cases. Decolonization, the goal of which is to decrease or eliminate bacterial load on the body, is an integral part of the strategies used to control and prevent the spread of MRSA. This approach involves eradication of MRSA carriage from the nose through the intranasal application of an antimicrobial agent and body washes with an antiseptic soap to eliminate bacteria from other body sites. The most commonly used agents for MRSA decolonization are intranasal mupirocin ointment applied to the anterior nares and chlorhexidine body wash. Postdischarge MRSA decolonization with chlorhexidine and mupirocin led to a 30% lower risk of MRSA infection. However, there are growing concerns about decolonization failures following the emergence of mupirocin and chlorhexidine resistance. Povidone iodine (PVP-I) is an alternative decolonization agent solutions and demonstrated rapid and superior bactericidal activity against MRSA in in vitro and ex vivo studies available reports. Finally, the induction of bacterial resistance or cross-resistance to antiseptics and antibiotics with PVP-I was not observed. The present protocol aims to use a "Decolonization kit" into MRSA patients to evaluate the efficacy of MRSA nasal decolonization with a topical PVP-I gel. This kit will allow a complete transient decolonization with povidone-iodine (PVP-I)-based products: nasal (gel), body (antiseptic soap) and oral (mouthwash).

ELIGIBILITY:
Inclusion Criteria:

* Patients readmitted at the Nantes University Hospital and detected to be already MRSA positive by nasal systematic screening,
* MRSA patients with length of hospital stay > 4 days
* Patient older than 18 years and informed about the study,
* Patients who provide their written informed consent,
* Patient affiliated with French social security system or beneficiary from such system.

Women must meet one of the following criteria at the time of inclusion:

* use adequate contraceptive measures as recommended by the CTFG (Recommendations related to contraception and pregnancy testing in clinical trials v1.1), and have a negative pregnancy test (urine test) prior to receiving the first dose of study drug;
* or be post-menopausal (over 50 years of age with amenorrhea for at least 12 months after discontinuation of all exogenous hormonal therapy)
* or (if under 50 years of age) have been amenorrheic for at least 12 months after discontinuation of exogenous hormonal therapy and with luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels corresponding to post-menopausal levels
* or have undergone irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy (this operation must be documented).

Exclusion Criteria:

* Patient < 18 years,
* Patient with known intolerance to PVD-I derivatives or excipients
* Known MRSA colonized patient managed in outpatient or inpatient care but with a negative nasal screen,
* New patient with MRSA infection (this patient can be included later in case of hospital readmission),
* Pregnancy or breastfeeding, patient with childbearing potential that refused acceptable contraceptive method
* Patients with a known risk of allergy to povidone iodine,
* Patients with damaged skin or mucous,
* Patients with a history of thyroid disorders,
* Adults under guardianship or trusteeship,
* Patients under juridical protection
* Use of mercurial antiseptic during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-11-21 (Actual); Primary Completion 2025-12-04 (Actual); Study Completion 2025-12-04 (Actual)

PRIMARY OUTCOMES:
MRSA nasal decolonization: Negative nasal screening rate 6 hours after use of the kit. | 6 hours

SECONDARY OUTCOMES:
Acceptability by the patient and HCWs of the use of the complete kit by a satisfactory self- questionnaire. | 24 hours
Characteristics of patients remained MRSA positive after PVP-I decolonization. | 24 hours
List of adverse events reported by patients. | 24 hours
MRSAD decolonization: negative nasal screening rate 24 hours after use of the kit | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No